CLINICAL TRIAL: NCT02564354
Title: Open-Label, Exploratory Study to Evaluate the Effects of QR-010 on Nasal Potential Difference in Subjects With CF With the ΔF508 CFTR Mutation
Brief Title: Exploratory Study to Evaluate QR-010 in Subjects With Cystic Fibrosis ΔF508 CFTR Mutation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ProQR Therapeutics (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PQ-010-002
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CF; ΔF508; CFTR; QR-010; antisense oligonucleotide; RNA therapy; F508del; NPD; nasal potential difference
MeSH Terms: conditions — Cystic Fibrosis | interventions — eluforsen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ΔF508 Homozygous (Experimental): QR-010 administered intranasally as an atomized liquid 10 mg (5 mg per nostril), 3 times weekly for 4 weeks.
  Interventions: Drug: QR-010
- ΔF508 Compound Heterozygous (Experimental): QR-010 administered intranasally as an atomized liquid 10 mg (5 mg per nostril), 3 times weekly for 4 weeks.
  Interventions: Drug: QR-010

INTERVENTIONS:
Drug: QR-010 — Single-stranded RNA antisense oligonucleotide in isoosmolar solution

SUMMARY:
Exploratory proof of concept study to determine whether intranasal administration of QR-010 in subjects with cystic fibrosis, homozygous or compound heterozygous for the ΔF508 mutation, can increase the function of Cystic Fibrosis Transmembrane Conductance Regulator (CFTR).

DETAILED DESCRIPTION:
This is an open-label, multi-center, exploratory study to estimate the effect of intranasal administration of QR-010 on the nasal mucosa in the restoration of CFTR function, as measured by nasal potential difference (NPD), in the nasal epithelium of adult subjects with CF who are homozygous or compound heterozygous for the ΔF508 CFTR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF as defined by iontophoretic pilocarpine sweat chloride test (sweat chloride) of > 60 mmol/L
* Nasal potential difference (NPD) measurement at Screening consistent with CF
* Confirmation of CFTR gene mutations homozygous or compound heterozygous for the ΔF508 mutation
* Body mass index (BMI) of ≥ 18 kg/m2
* Non-smoking for a minimum of 2 years
* Stable lung function
* FEV1 ≥40% of predicted normal for age, gender, and height at Screening

Exclusion Criteria:

* Breast-feeding or pregnant
* Acute allergy or infection affecting nasal conditions not resolved within 14 days prior Screening
* Use of lumacaftor or ivacaftor
* Use of any investigational drug or device
* Hemoptysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Clancy, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (5):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - National Jewish Health, Denver, Colorado
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
- U.Z. Leuven, Leuven, Belgium
- Hopital Necker-Enfants Malades, Paris, France

REFERENCES:
- [Derived] Miah KM, Hyde SC, Gill DR. Emerging gene therapies for cystic fibrosis. Expert Rev Respir Med. 2019 Aug;13(8):709-725. doi: 10.1080/17476348.2019.1634547. Epub 2019 Jun 27. PMID 31215818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 5 hospitals in the USA and Europe. Screenings for Cohort 1 and Cohort 2 occurred in parallel between between 19th October 2015 and 14th July 2016.
Groups:
- Cohort 1: Homozygous for the F508del-CFTR Mutation: Subjects homozygous for the F508del-CFTR (Cystic Fibrosis Transmembrane conductance Regulator) mutation were enrolled into Cohort 1 and received QR-010 10 mg (5 mg/250 μL saline per nostril) via bilateral intranasal administration three times a week for 4 weeks for a total of 12 doses.
- Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation: Subjects compound heterozygous for the F508del-CFTR mutation were enrolled into Cohort 2 and received QR-010 10 mg (5 mg/250 μL saline per nostril) via bilateral intranasal administration three times a week for 4 weeks for a total of 12 doses.
Period: Overall Study
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Homozygous for the F508del-CFTR Mutation: Subjects homozygous for the F508del-CFTR mutation were enrolled into Cohort 1 and received QR-010 10 mg (5 mg/250 μL saline per nostril) via bilateral intranasal administration three times a week for 4 weeks for a total of 12 doses.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 25.80 [19 to 36] | 36.00 [18 to 63] | 30.33 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 4 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 2 | 2 | 4
  United States | 4 | 5 | 9
  France | 4 | 1 | 5
FEV1% predicted [Mean (Full Range); unit: Percent of the predicted value] — Lung function; Forced Expiratory Volume in 1 second; a percent of the "predicted values" of patients with similar characteristics.
  Percent of the predicted value | 74.22 [45.16 to 108.77] | 73.55 [52.25 to 93.80] | 73.92 [45.16 to 108.77]

OUTCOME MEASURES:

1. Primary Outcome: Intra-subject Change From Baseline of CFTR-mediated Total Chloride Transport as Measured by Nasal Potential Difference (NPD).
Description: The primary endpoint was the within-subject change from baseline in total chloride transport as measured by NPD, after the Chloride-free+isoproterenol solution (Cl-free+iso), and was based on the average measurements of both nostrils. To provide baseline stability, baseline was defined as the average of the two most recent pre-dose values, where each pre-dose value was the average of two nostrils. A negative change from baseline of Cl-free+iso shows an improvement.
Time Frame: Baseline, at 2 and 4 weeks, and at 3 weeks post-treatment.
Population: Per Protocol Set: 3 subjects from Cohort 1 and 1 subject from Cohort 2 didn't meet the NPD entry criterion and were excluded from the per protocol analysis. Further 1 subject from Cohort 1 did not have an interpretable Week 4 NPD measurement.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Number analyzed (Participants) | 7 | 7
mV
  Baseline | 1.86 (3.360) | -0.75 (3.868)
  Week 2 | -1.11 (8.062) | 1.66 (3.937)
  Week 4: number analyzed (Participants) | 6 | 7
  Week 4 | -1.92 (4.837) | 1.43 (2.644)
  3 weeks post-treatment | -1.86 (6.736) | 2.27 (6.546)

2. Secondary Outcome: Number of Subjects With a -6.6 mV or More Negative Change in CFTR-mediated Total Chloride Transport, and After Different Treatment Durations From Baseline Through End of Study.
Description: This analysis is the proportion (amount) of subjects with an average Cl-free+iso actual value of -6.6 mV or more negative after treatment (ie, responders), as measured by NPD and was based on the average measurements of both nostrils. The actual value of -6.6 mV is used to discriminate individuals with CF (>-6.6 mV) from normal individuals (≤ -6.6 mV).
Time Frame: 2 and 4 weeks, and at 3 weeks post-treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Number analyzed (Participants) | 7 | 7
Participants
  Week 2 | 1 | 0
  Week 4: number analyzed (Participants) | 6 | 7
  Week 4 | 1 | 0
  3 weeks post-treatment | 2 | 0

3. Secondary Outcome: Number of Subjects With a -4 mV or More Negative Change in CFTR-mediated Total Chloride Transport, and After Different Treatment Durations From Baseline Through End of Study.
Description: This analysis is the proportion of subjects with an average Cl-free+iso actual value of -4 mV or more negative after treatment (ie, responders), as measured by NPD and was based on the average measurements of both nostrils. The value of -4 mV is considered a clinically relevant response to treatment based on data from studies of other CFTR therapies.
Time Frame: 2 and 4 weeks, and at 3 weeks post-treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Number analyzed (Participants) | 7 | 7
Participants
  Week 2 | 3 | 1
  Week 4: number analyzed (Participants) | 6 | 7
  Week 4 | 2 | 1
  3 weeks post-treatment | 4 | 0

4. Secondary Outcome: Intra-subject Change of Sodium Transport as Measured by Nasal Potential Difference (NPD) From Baseline Through End of Study.
Description: This endpoint was the within-subject change in Sodium transport (average Potential Difference prior to perfusion of any solution); this is the average of Potential Difference measured at five sites in the inferior meatus of the nose. A positive change from baseline shows an improvement.
Time Frame: Baseline, at 2 and 4 weeks, and at 3 weeks post-treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Number analyzed (Participants) | 7 | 7
mV
  Baseline | -31.92 (8.777) | -27.02 (11.412)
  Week 2 | -33.80 (9.922) | -27.48 (9.230)
  Week 4: number analyzed (Participants) | 6 | 7
  Week 4 | -25.14 (10.809) | -25.52 (10.445)
  3 weeks post-treatment | -31.56 (7.791) | -27.59 (6.291)

5. Secondary Outcome: The Mean Change in CFTR-mediated Total Chloride Transport.
Description: The mean change in CFTR-mediated Total Chloride Transport compared to Baseline, per cohort; this is the mean of Potential Difference measured at five sites in the inferior meatus of the nose measured in millivolts (mV). A negative change from baseline shows an improvement.
Time Frame: 2 and 4 weeks, and at 3 weeks post-treatment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mV
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Number analyzed (Participants) | 7 | 7
mV
  Week 2 | -2.44 (2.00) | 1.88 (2.00)
  Week 4: number analyzed (Participants) | 6 | 7
  Week 4 | -3.46 (1.88) | 1.65 (1.70)
  3 weeks post-treatment | -3.19 (2.26) | 2.49 (2.26)

6. Secondary Outcome: Number of Subjects Experiencing Serious Adverse Events From Baseline Through End of Study.
Description: Number of subjects experiencing serious adverse events from baseline through End of Study.
Time Frame: 3 weeks post-treatment.
Population: Safety population: all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Number analyzed (Participants) | 10 | 8
Participants | 0 | 0

7. Secondary Outcome: Number of Subject Discontinuations Due to AEs From Baseline Through End of Study.
Description: Number of subject discontinuations due to AEs from baseline through End of Study. No discontinuations occurred.
Time Frame: 3 weeks post-treatment.
Population: Safety population: all subjects enrolled in the study; incidence of discontinuations due to AEs from baseline through End of Study will be reported in the Adverse Events section. No discontinuations occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Number analyzed (Participants) | 10 | 8
Participants | 0 | 0

8. Secondary Outcome: Number of Subjects With Abnormalities of Laboratory Parameters From Baseline Through End of Study.
Description: Number of subjects experiencing at least one abnormality in laboratory parameters (chemistry, hematology and urinalysis) that were reported as treatment emergent adverse event with a relationship to study drug as either possibly, probably or definitely, from baseline through End of Study.
Time Frame: 3 weeks post-treatment.
Population: Safety population: all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Number analyzed (Participants) | 10 | 8
Participants | 0 | 0

9. Secondary Outcome: Number of Subjects With Abnormalities of Vital Signs & Oximetry From Baseline Through End of Study.
Description: Number of subjects experiencing at least one abnormality vital signs & oximetry that were reported as treatment emergent adverse event with a relationship to study drug as either possibly, probably or definitely, from baseline through End of Study.
Time Frame: 3 weeks post-treatment.
Population: Safety population: all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Number analyzed (Participants) | 10 | 8
Participants | 0 | 0

10. Secondary Outcome: Number of Subjects With Abnormalities of Physical Examinations From Baseline Through End of Study.
Description: Number of subjects experiencing at least one abnormality in physical examination that were reported as treatment emergent adverse event with a relationship to study drug as either possibly, probably or definitely, from baseline through End of Study.
Time Frame: 3 weeks post-treatment.
Population: Safety population: all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Number analyzed (Participants) | 10 | 8
Participants | 3 | 4

11. Secondary Outcome: Changes in Nasal Symptoms (Based on the Nasal Examination Rating Scale - NERS) From Baseline Through End of Study.
Description: The NERS was performed by site staff prior to each dose and as part of the NPD procedure; it is a set of scales ranging from 0 (no symptoms) to 3 (most severe symptoms) for assessing the severity of each of the following nasal symptoms, separately for each nostril: mucosal disruption, edema, erythema, polyp, secretions. The range of the total sum is 0-30.
Time Frame: 3 weeks post-treatment.
Population: Safety population: all subjects enrolled in the study. 1 measurement was missing from 1 subject in Cohort 2 for Week 4.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Number analyzed (Participants) | 10 | 8
units on a scale
  Baseline | 12.20 (1.317) | 11.50 (1.773)
  Day 3 | 11.60 (1.647) | 13.38 (3.335)
  Day 5 | 11.50 (1.650) | 12.25 (2.550)
  Week 1 | 12.60 (2.171) | 12.00 (1.852)
  Day 10 | 11.50 (1.900) | 11.88 (2.532)
  Day 12 | 11.50 (1.269) | 11.50 (1.414)
  Week 2 | 12.50 (2.635) | 11.75 (1.909)
  Day 17 | 11.20 (2.098) | 12.00 (2.878)
  Day 19 | 11.90 (2.183) | 11.63 (1.923)
  Week 3 | 13.10 (2.685) | 12.63 (2.134)
  Day 24 | 11.90 (2.378) | 12.38 (2.326)
  Week 4: number analyzed (Participants) | 10 | 7
  Week 4 | 13.00 (2.828) | 11.71 (1.890)
  3 weeks post-treatment | 12.30 (2.541) | 12.75 (3.327)

12. Secondary Outcome: Changes in Nasal Symptoms (Sino-Nasal Outcome Test - SNOT-22) From Baseline Through End of Study.
Description: Subjects were asked to score a list of 22 symptoms on the SNOT-22 regarding social and emotional consequences. Outcomes were graded as 0 (no problem), to 5 (problem as bad as it could be). The list included: need to blow nose, sneezing, dripping nose, cough, postnasal drip, dense nasal drip, ear fullness, dizziness, ear pain, facial pain/pressure, difficulty falling asleep, waking at night, lack of a good night's sleep, waking up tired, fatigue, reduced productivity, reduced concentration, frustrated/restless/irritable, sad, embarrassed, decrease in smell and taste, and nasal obstruction. The range of the total sum is 0-110, with higher values indicating worse outcome.
Time Frame: 3 weeks post-treatment.
Population: Safety population: all subjects enrolled in the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
Number analyzed (Participants) | 10 | 8
units on a scale
  Baseline | 14.90 (5.896) | 19.13 (17.707)
  Week 2 | 13.60 (8.369) | 15.38 (18.601)
  Week 4 | 14.50 (11.048) | 14.13 (16.084)
  3 weeks post-treatment | 10.70 (8.301) | 14.50 (10.915)

ADVERSE EVENTS:
Time Frame: After the subject had provided informed consent, but prior to initiation of IMP, only SAEs caused by a protocol-mandated intervention were collected. After initiation of IMP, all AEs and SAEs, regardless of attribution, were collected until at least 30 days following the last administration of IMP or initiation of new therapy, whichever was earlier.
Arm/Group | Cohort 1: Homozygous for the F508del-CFTR Mutation | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 9/10 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Homozygous for the F508del-CFTR Mutation (N=10) | Cohort 2: Compound Heterozygous for the F508del-CFTR Mutation (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 4
Malaise (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Galbladder pain (Hepatobiliary disorders) | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 3 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intranasal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal mucosal erosion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators are restricted from disclosure or results until after multi-center publication or 12 months after the completion of the Study at all participating research centers. Sponsor can review results communication prior to public release and can embargo communications regarding trial results for a period that is more than 60 days (varying per site). Sponsor may request redaction of confidential information.